The Impact of Semaglutide on Gut Microbiota in Obese Patients

Research Unit: Beijing Chaoyang Hospital, Capital Medical University

Principal Investigator: Jia Liu

1. Research Background and Rationale

Obesity is a chronic disease characterized by excessive fat deposition, which increases

the risk of hypertension, diabetes, non-alcoholic fatty liver disease, sleep apnea

syndrome, coronary heart disease, and other conditions. Ultimately, it affects patients'

life expectancy and raises healthcare costs, making it one of the most severe global

public health issues [1]. Weight loss can significantly reduce the risk of

obesity-related complications [2]. Lifestyle interventions are the first-line treatment

for obesity management, but even with strict adherence, they typically result in only a

5–10% reduction in body weight, which is difficult to maintain long-term. There is an

urgent need for the development of highly effective and safe weight-loss drugs.

Glucagon-like peptide-1 (GLP-1) receptor agonists, represented by semaglutide, have

been approved for chronic weight management in obese patients [6–7]. Numerous

studies have shown that semaglutide treatment significantly reduces body weight in

obese patients with a good safety profile [7]. However, it is noteworthy that the

weight-loss effects of semaglutide exhibit significant individual variability [4–5]. The

STEP-5 trial found that semaglutide treatment resulted in an average weight loss of

15.2% in non-diabetic obese or overweight adults, but 23% of participants showed no

significant weight reduction [4]. The recently published SELECT trial revealed that

32.2% of obese or overweight adults experienced no significant weight changes after

using semaglutide [5].

The gut microbiota plays a crucial role in maintaining host physiology and

homeostasis [8]. Our previous research demonstrated that metformin treatment

reduces the abundance of Bacteroides fragilis and increases levels of

glycoursodeoxycholic acid (GUDCA), thereby improving blood glucose and insulin

resistance [9]. Time-restricted feeding was found to increase the abundance

of Ruminococcus torques (R. torques), which produces 2-hydroxy-4-methylpentanoic

acid (HMP) to inhibit the intestinal hypoxia-inducible factor- $2\alpha$  (HIF- $2\alpha$ )-ceramide

pathway, thereby ameliorating liver inflammation and fibrosis in mice [10]. Recent

studies have shown that gut microbiota also modulates host responses to treatments,

contributing to individual variability in drug efficacy [11]. J. Balaich et al. discovered

that microbial-derived acarbose kinases specifically metabolize and deactivate

acarbose, affecting its glucose-lowering effects [12]. Our team previously found that

gut microbial dipeptidyl peptidase-4 (DPP4) enters intestinal tissues under conditions

of intestinal barrier damage, degrading active host GLP-1 and inducing glucose

intolerance. Host DPP4 inhibitors like sitagliptin cannot effectively inhibit microbial

DPP4 activity, which is a major reason for the high variability in clinical responses to

sitagliptin [13].

In our preliminary study, we performed fecal metagenomic sequencing on obese

patients treated with semaglutide, matched for baseline gender, age, and body mass

index (BMI), and observed significant differences in gut microbiota composition and

abundance before and after treatment. Further experiments in a high-fat diet-induced

obese mouse model revealed that antibiotic treatment enhanced the weight-loss effects

of semaglutide. These findings suggest that gut microbiota modulates host responses

to semaglutide treatment, although the specific mechanisms remain unclear.

This study aims to elucidate the impact of semaglutide on gut microbiota in obese

patients and explore the development of targeted microbial enzyme therapies,

providing new targets for overcoming semaglutide resistance in weight loss.

2. Research Objectives

This study will employ fecal metagenomic sequencing and multi-omics technologies,

along with an in vitro bacterial strain screening platform, to investigate the effects of

semaglutide on gut microbiota in obese patients and elucidate the underlying

mechanisms. The goal is to identify novel targets for developing drugs to overcome

semaglutide resistance in weight loss.

3. Research Methods

3.1 Study Setting and Population

Obese patients visiting the Department of Endocrinology at Beijing Chaoyang

Version Number: V2.0

Hospital, Capital Medical University, from April 2025 to April 2026 will be recruited based on the following inclusion and exclusion criteria:

#### Inclusion Criteria:

- Age 18–60 years;
- BMI  $\geq$  30 kg/m<sup>2</sup>;
- At least one self-reported unsuccessful attempt at lifestyle-based weight loss;
- Willingness to participate and signed informed consent.

### **Exclusion Criteria:**

- Self-reported weight change >5% in the 3 months before screening;
- Use of any weight-loss medication in the 3 months before screening;
- Use of glucose-lowering drugs in the 3 months before screening, HbA1c ≥ 6.5%, or history of type 1 or type 2 diabetes;
- Use of immunosuppressants, steroids, antidiarrheals, antibiotics, probiotics, lipid-lowering drugs, or other gastrointestinal motility drugs in the 3 months before screening;
- History of endocrine-related overweight or obesity (e.g., Cushing's syndrome);
- Triglycerides ≥500 mg/dL (5.65 mmol/L) at screening;
- Clinically significant gastric emptying abnormalities (e.g., severe diabetic gastroparesis or gastric outlet obstruction), gastrointestinal diseases, or surgical history;
- Thyroid dysfunction;
- History of mental illness;
- Personal or family history of multiple endocrine neoplasia or medullary thyroid carcinoma, or calcitonin ≥6 pg/mL;
- Abnormal liver function at screening (ALT and/or AST >3× ULN);
- Abnormal renal function at screening (eGFR <60 mL/min/1.73 m<sup>2</sup>);
- History of cardiovascular disease;
- History of malignancy;
- Pregnancy or lactation;
- Other conditions deemed unsuitable for participation by the investigator.

3.2 Study Design

Recruitment:

A self-controlled cohort study design will be used to recruit obese patients from the

Department of Endocrinology at Beijing Chaoyang Hospital from April 2025 to April

2026.

Treatment and Follow-up:

Eligible participants will receive subcutaneous semaglutide injections. The treatment

follows a dose-escalation regimen to achieve steady-state plasma concentrations over

4–5 weeks: Start with 0.5 mg once weekly; Increase to 1.0 mg once weekly after 4

weeks; Further increase to 1.7 mg once weekly after another 4 weeks; Total treatment

duration: 12 weeks.

Participants will visit the clinic every 4 weeks for follow-up assessments, including

general condition, physical examinations, and laboratory tests. At the 12-week

follow-up, venous blood will be collected for semaglutide plasma concentration

analysis.

Outcome Measures:

Primary Outcome: Changes in gut microbiota composition (abundance and Shannon

diversity index) from baseline to 12 weeks.

Secondary Outcomes: Changes in weight, BMI, waist circumference, hip

circumference, and lipid profiles from baseline to 12 weeks.

3.3 Sample Size Calculation

A paired t-test will be used for pre-post comparisons. Based on prior studies, the

standard deviation of paired differences ( $\sigma$ d) is 1.2, the clinically meaningful minimal

difference ( $\Delta$ ) is 1.0,  $\alpha = 0.05$  (two-tailed),  $Z_1 - \alpha/2 = 1.96$ ,  $\beta = 0.1$  (Power = 90%),

and  $Z_1$  - $\beta$  = 1.28. The calculated sample size is 16, accounting for a 20% dropout rate

and 30% redundancy in microbiome data. The final sample size is 40, with

adjustments based on recruitment feasibility.

3.4 Data Collection

1) Anthropometric Data:

Height, weight, BMI, waist/hip circumference, blood pressure, etc., measured by

Version Number: V2.0

trained staff.

2) Urine and Fecal Samples:

Urine: Midstream samples collected for biochemical analysis and stored at -80°C.

Fecal: Fresh samples collected internally to avoid contamination, stored at -80°C for metagenomic sequencing. DNA extraction, sequencing (Illumina HiSeq 4000), and

bioinformatics analysis will be performed.

3) Blood Samples:

Fasting venous blood for routine tests (glucose, insulin, HbA1c, lipids, etc.) and semaglutide concentration (LC-MS/MS).

3.5 Follow-up Schedule

Participants will be followed every 4 weeks for 12 weeks, with assessments including physical exams, lab tests, and safety monitoring.

3.6 Data Management and Statistical Analysis

Data Management:

Double-entry verification using Epidata, with logic checks and error correction before database locking.

Statistical Analysis:

SPSS for analysis.

Normal distribution: Mean  $\pm$  SD (paired t-test); non-normal: Median (IQR) (Wilcoxon test).P < 0.05 considered statistically significant.

3.7 Bias Control

Strict adherence to inclusion/exclusion criteria, standardized data collection, and multivariate regression to adjust for confounders (age, sex, baseline BMI, diet).

4. Quality Control

Fecal sample collection: Avoid urine contamination, use sterile containers, store at -80°C.

Questionnaire integrity: Trained staff, regular audits.

Accurate measurements: Certified professionals, quality-controlled lab procedures.

5. Risk Assessment and Mitigation

Risks:

Blood draw: Syncope/hypoglycemia.

Semaglutide: GI discomfort, allergies.

Mitigation:

Emergency protocols for adverse events.

Dose escalation and monitoring to minimize risks.

# **6. Expected Outcomes**

Elucidate semaglutide's impact on gut microbiota and mechanisms.

Identify targets for overcoming resistance.

Publish 2–3 high-impact papers; patent applications if biomarkers are discovered.

#### 7. Timeline

Period Tasks

2025.04–2025.09 Recruitment and follow-up

2025.10–2025.12 Data analysis

2026.01–2026.04 Manuscript preparation/submission

## References

- 1. Gilden AH, Catenacci VA, Taormina JM. The Obesity. Ann Intern Med. 2024.
- 2. Tahrani A, Morton J. Benefits of weight loss of 10% or more in patients with overweight or obesity: A review. Obesity. 2022;30(4):802-840.
- 3. Papamargaritis D, le Roux CW, Holst JJ, Davies MJ. New therapies for obesity. Cardiovasc Res. 2024;119(18):2825-2842.
- 4. Garvey WT, Batterham RL, Bhatta M, Buscemi S, Christensen LN, Frias JP, Jódar E, Kandler K, Rigas G, Wadden TA, Wharton S, Grp SS. Two-year effects of semaglutide in adults with overweight or obesity: the STEP 5 trial. Nat Med. 2022;28(10):2083-2091.
- 5. Ryan DH, Lingvay I, Deanfield J, Kahn SE, Barros E, Burguera B, Colhoun HM, Cercato C, Dicker D, Horn DB, Hovingh GK, Jeppesen OK, Kokkinos A, Lincoff AM, Meyhöfer SM, Oral TK, Plutzky J, van Beek AP, Wilding JPH, Kushner RF. Long-term weight loss effects of semaglutide in obesity without diabetes in the SELECT trial. Nat Med. 2024.
- 6. Moore PW, Malone K, VanValkenburg D, Rando LL, Williams BC, Matejowsky HG, Ahmadzadeh S, Shekoohi S, Cornett EM, Kaye AD. GLP-1 Agonists for Weight Loss: Pharmacology and Clinical Implications. Adv Ther. 2023;40(3):723-742.

- 7. Moiz A, Levett JY, Filion KB, Peri K, Reynier P, Eisenberg MJ. Long-Term Efficacy and Safety of Once-Weekly Semaglutide for Weight Loss in Patients Without Diabetes: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Am J Cardiol. 2024;222:121-130.
- 8. Busch CBE, Bergman JJGHM, Nieuwdorp M, van Baar ACG. Role of the Intestine and Its Gut Microbiota in Metabolic Syndrome and Obesity. Am J Gastroenterol. 2024;119(6):1038-1046.
- 9. Sun LL, Xie C, Wang G, Wu Y, Wu Q, Wang XM, Liu J, Deng YY, Xia JL, Chen B, Zhang SY, Yun CY, Lian G, Zhang XJ, Zhang H, Bisson WH, Shi JM, Gao XX, Ge PP, Liu CH, Krausz KW, Nichols RG, Cai JW, Rimal B, Patterson AD, Wang X, Gonzalez FJ, Jiang CT. Gut microbiota and intestinal FXR mediate the clinical benefits of metformin. Nat Med. 2018;24(12):1919-1929.
- 10. Zhang, Y., Wang, X., Lin, J., Liu, J., Wang, K., Nie, Q., Ye, C., Sun, L., Ma, Y., Qu, R., Mao, Y., Zhang, X., Lu, H., Xia, P., Zhao, D., Wang, G., Zhang, Z., Fu, W., Jiang, C., & Pang, Y. (2024). A microbial metabolite inhibits the HIF-2α-ceramide pathway to mediate the beneficial effects of time-restricted feeding on MASH. Cell metabolism, 36(8), 1823–1838.e6.
- 11. Javdan B, Lopez JG, Chankhamjon P, Lee YCJ, Hull R, Wu QH, Wang XJ, Chatterjee S, Donia MS. Personalized Mapping of Drug Metabolism by the Human Gut Microbiome. Cell. 2020;181(7):1661-1679.
- 12. Balaich J, Estrella M, Wu GJ, Jeffrey PD, Biswas A, Zhao LP, Korennykh A, Donia MS. The human microbiome encodes resistance to the antidiabetic drug acarbose. Nature. 2021;600(7887):110-115.
- 13. Wang K#, Zhang ZW#, Hang J#, Liu J#, Guo FS#, Ding Y, Li M, Nie QX, Lin J, Zhuo YY, Sun LL, Luo X, Zhong QH, Ye C, Yun CY, Zhang Y, Wang J, Bao R, Pang YL, Wang G\*, Gonzalez FJ\*, Lei XG\*, Qiao J\*, Jiang CT\*. Microbial-host-isozyme analyses reveal microbial DPP4 as a potential antidiabetic target. Science. 2023;381(6657):eadd5787.